CLINICAL TRIAL: NCT05733325
Title: Diet-induced Elevations in LDL-C and Progression of Atherosclerosis
Acronym: Keto-CTA
Status: Completed | Type: Observational
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Collaborators: Citizen Science Foundation (Unknown)
Responsible Party: Principal Investigator, Matthew J. Budoff, Professor of Medicine, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Other Study IDs: CSF-A1
Record Dates: First submitted 2023-02-08; First posted 2023-02-17 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational study examining the progression of subclinical coronary atherosclerosis in healthy participants who have an elevated LDL-C (above 190mg/dl) secondary to diet not associated with genetic familial hypercholesterolemia (FH). This study participants are classified to be Lean-Mass-Hyper-Responder (LMHR).

DETAILED DESCRIPTION:
This is an observational study examining the progression of subclinical coronary atherosclerosis in healthy participants who have an elevated LDL-C (above 190mg/dl) secondary to diet not associated with genetic familial hypercholesterolemia (FH). The investigator proposes to measure subclinical atherosclerosis as measured by low-dose prospective ECG-triggered cardiac computed tomographic angiography (CCTA) - in order to evaluate the rates of progression of atherosclerosis over 1 year. These participants will have voluntarily been eating a very low carbohydrate or ketogenic diet (VLC/KD) for at least 24 months, with evidence of significant elevations in LDL-C after commencing the diet.

Participants will be recruited online through social media including Facebook groups discussing VLC/KDs. The target population are those who experience significant increases in LDL-C on VLC/KDs whilst also being healthy and relatively lean (BMI <30mg/kg2 and waist circumference <102 cm and 88 cm for men and women respectively if BMI 25-30 mg/kg2).

Once participants present their interest to participate in the study by responding to the social media flyer and made an attempt to get in touch with the study site, study staff will reach out to the participant over the phone using an IRB (Institutional Review Board) approved screening questionnaire to verify eligibility and answer any question about the study. Once subject confirms that he/she is interested to participate, they will be informed that a copy of the Informed Consent Form (ICF) will be emailed to them using a HIPAA compliant DocuSign (application to sign a document electronically) portal. Subjects are required to review and electronically sign the ICF. Once an ICF has been signed, subject will be asked to upload the relevant medical records to the HIPAA compliant RedCap portal as documentary evidence to the lipid levels. Once the study team reviews the medical records/lab results and confirm the subject eligibility, the travel arrangements to the study site for the in-person baseline visit will be made.

Study participants will have total of 2 in-person study visits (Baseline - visit 1 and 12 month - visit 2) and will have a 6 month - phone visit in between.

During the baseline site visit, the participants will be asked to take a genetic test, blood draw, ECG and CCTA. Study staff will also be collecting vital signs, medical history, physical exam and questionnaire. Study participants will be asked to measure their morning blood ketone and glucose levels every day and report the results using KetoMojo application.

Subjects will be informed about the possible risk associated with the study participation including radiation from the CT scan/CCTA, risks associated with the taking Beta-blocker, Calcium channel blocker, Nitroglycerin as well as IV insertion.

Recruitment will take place over 6 months, with follow up over 12 months. The study design calls for the enrollment of 100 eligible subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Had an LDL cholesterol of 160 mg/dL or below from most recent labs taken before adopting a low carb diet (requires documentary evidence)
* Has seen an increase of LDL cholesterol to 190 mg/dL or above from most recent labs on current diet **
* Has LDL cholesterol levels at least 50% or greater compared to most recent documented value prior to starting the diet.
* On low carb, ketogenic diet for the last 24 months or more.
* HDL-C ≥ 60 mg/dL and triglyceride level ≤ 80 mg/dL **
* Willingness to participate in the study and ability to sign informed consent
* In the investigator's opinion subjects are willing and likely able to comply with scheduled visits, laboratory tests, and other study procedures.
* Normal to low BP (systolic ≤ 130 mm Hg or diastolic ≤ 80 mm Hg) at screening/baseline (visit 1).
* Fasting glucose < 110 mg/dL and HbA1c < 6.0%) **
* hsCRP < 2 mg/L **
* No prior diagnosis of Type 2 Diabetes
* No prior use of anti-diabetic medication
* Not currently taking lipid lowering supplements or medications including statins, red yeast rice, garlic, ezetimibe, berberine

  * Requires documentary evidence

Exclusion Criteria:

* Untreated hypothyroidism (TSH > 10)
* Use of medications that elevated LDL-C (anabolic steroids, isotretinoin, immunosuppressants, amiodarone, thiazide diuretics, glucocorticoids, or thiazolidinediones)
* Pregnancy
* Has smoked more than 100 cigarettes in lifetime
* An ongoing inflammatory disorder (e.g. psoriatic arthritis)
* History of atherosclerotic heart disease
* Known history of molecularly defined Familial Hypercholesterolemia
* BMI = or > 30 kg/m^2 (or waist circumference > 88 cm or > 102 cm for women and men respectively if BMI between 25-30 kg/m^2)
* Renal insufficiency (calculated creatinine clearance of <50 ml per minute, MDRD (modification of Diet in Renal Disease) equation).
* Use of Lipid lowering medication (Statins, etc) at the time of most recent labs taken before starting Ketogenic diet.
* AST (Aspartate aminotransferase) or ALT (Alanine Transaminase) >2 times the upper limit of normal (ULN) at the Screening visit (V1), or a total bilirubin >1.5 times the ULN unless the subject has a history of Gilbert's.
* Subject unable to provide medical records indicating lab results before starting a keto- diet.
* Subject has a history of malignancy ≤5 years prior to signing informed consent, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer.
* Note (1) A subject with a history of malignancy >5 years prior to signing informed consent should have no evidence of residual or recurrent disease.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality at the Screening visit (V1) that may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of trial results and, in the judgment of the investigator, would make the subject inappropriate for entry into this trial.
* Subjects with known allergy to iodinated contrast material
* Subject is pregnant or breast-feeding, or is expecting to conceive during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Lean Mass Hyper-Responders: The target population are those who experience significant increases in LDL-C on VLC/KDs whilst also being healthy and relatively lean (BMI <30mg/kg2 and waist circumference <102 cm and 88 cm for men and women respectively if BMI 25-30 mg/kg2). These individuals are referred to as lean mass hyper-responders (LMHRs) with diet-induced hypercholesterolemia (DIH).
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2024-02-12 (Actual); Study Completion 2024-02-12 (Actual)

PRIMARY OUTCOMES:
Percent change in total non-calcified coronary plaque volume | 12 months
  Percent change in total non-calcified coronary plaque volume from baseline (start of the study) till the final visit will be measured using Coronary Computed Tomography Angiography (CCTA).

CONTACTS AND LOCATIONS:
Overall Officials: Matthew A Budoff, MD, Principal Investigator — The Lundquist Institute for Biomedical Innovation at Harbor UCLA Medical Center
Locations (1):
- Lundquist Institute for Biomedical Innovation at Harbor UCLA Medical Center (The Lundquist Institute), Torrance, California, United States

REFERENCES:
- [Derived] Soto-Mota A, Norwitz NG, Manubolu VS, Kinninger A, Wood TR, Earls J, Feldman D, Budoff M. Longitudinal Data From the KETO-CTA Study: Plaque Predicts Plaque, ApoB Does Not. JACC Adv. 2025 Jul;4(7):101686. doi: 10.1016/j.jacadv.2025.101686. Epub 2025 Apr 7. PMID 40192608